CLINICAL TRIAL: NCT00457314
Title: Exercise Training and Deconditions: Implications for Therapy in Mitochondrial Myopathy
Brief Title: The Effects of Exercise Versus Inactivity on People With Mitochondrial Muscle Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Ronald Haller, Universit y of Texas Southwestern Medical School
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R01AR050597 (NIH); 1R01AR050597-01A1 (NIH)
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Mitochondrial Myopathy
Keywords: single-large scale deletions; point mutations in mtDNA
MeSH Terms: conditions — Mitochondrial Myopathies | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will partake in regular exercise training for 6 months. After 6 months, they will switch to no exercise training for 6 months. Participants will then be encouraged to continue exercise training for an additional 1 year.
  Interventions: Behavioral: Exercise
- 2 (Experimental): Participants will not partake in regular exercise training for 6 months. After 6 months, they will switch to exercise training for 6 months. Participants will then be encouraged to continue exercise training for an additional 1 year.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Regular exercise training

SUMMARY:
Mitochondrial myopathies include various inherited diseases that are caused by damage to the mitochondria, energy-producing structures that fuel the body's processes. The main symptoms are muscle weakness, reduced muscle mass, and difficulty with exercising. The purpose of this study is to determine the effects of exercise training versus inactivity on mitochondrial function in muscle and muscle performance in people with mitochondrial myopathies.

DETAILED DESCRIPTION:
Mitochondrial myopathies are caused by mutant mitochondrial DNA, genetic defects in parts of the mitochondrial DNA. These defects can include missing or deleted DNA that typically codes for certain proteins involved in energy production. These mutations cause individual mitochondria and the body on a whole to produce energy less efficiently. Because muscle cells require extensive energy to function properly, they are particularly impaired by mitochondrial dysfunction. The onset of most mitochondrial myopathies occurs before the age of 20. Initially a person may experience muscle weakness and fatigue during physical activity. Other symptoms may include limited eye mobility, heart arrhythmias, slurred speech, swallowing difficulties, and impaired movement.

There is no cure yet for mitochondrial myopathies, nor is there any adequate treatment to stall disease progression. Exercise, known to boost the production and function of mitochondria in healthy people, may reduce symptoms in people with mitochondrial myopathies by increasing the number and function of normal mitochondria in an individual muscle cell. The purpose of this study is to determine the effects of exercise training versus inactivity on the expression of normal and mutant mitochondrial DNA and on mitochondrial production within muscle cells in people with mitochondrial myopathies. The study will also assess how cell function, physical endurance, heart function, and quality of life are affected by exercise training and inactivity.

Participants in this 2-year study will first undergo physiological exercise testing, magnetic resonance imaging (MRI) of heart and skeletal muscles, a needle biopsy of muscle, and a questionnaire on quality of life. Participants will then be randomly assigned to partake in regular exercise training or no training for 6 months. After 6 months, all participants will undergo repeat testing of initial evaluations. Participants who had been in the exercising group will then switch to no exercise training for 6 months, and participants who had been in the non-exercising group will switch to regular exercise training for 6 months. The second 6-month period will also be followed by repeat testing of initial evaluations. Participants will then be encouraged to continue exercise training for an additional 1 year, with retesting at the end of the second year. Each of the four evaluations will take about 15 hours over 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mitochondrial myopathy
* Single-large scale deletions of mitochondrial DNA
* Point mutations in mitochondrial DNA

Exclusion Criteria:

* Symptoms or electrocardiogram-generated signs of coronary artery disease
* Symptoms of congestive heart failure; peripheral vascular disease; or lung, kidney, or liver disease
* History of alcohol or substance abuse
* Metal implants or related devices that contraindicate MRI
* Current use of or require any medications that have significant systemic cardiovascular effects
* Diabetes
* Obesity (body mass index [BMI] greater than 30)
* Resting systolic blood pressure greater than 140 mmHg and/or diastolic blood pressure greater than 90 mmHg at three different times

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Changes in wild-type (normal), mutant, and total mitochondrial DNA copy number | Measured at Week 26
Physiological measure of oxidative metabolism | Measured at Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Haller, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States